CLINICAL TRIAL: NCT06608849
Title: A Non-interventional, Prospective, Cross-sectional Study of the Incidence of Pulmonary, Cardiovascular and Renal System Non-communicable Complications Associated With the Post-acute Phase of the Infection by Sars-Cov-2
Brief Title: The Incidence of Pulmonary, Cardiovascular and Renal System Non-communicable Complications Associated With the Post-acute Phase of the Infection by Covid-19
Acronym: POINT
Status: Recruiting | Type: Observational
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Other Study IDs: POINT
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Complications; Cardiovascular Complications; Renal Complications; COVID-19
Keywords: Covid-19; SARS-CoV-2; Pulmonary complications; Cardiovascular complications; Renal complications; Post-acute phase; Non communicable diseases; Biomarkers; Prevention
MeSH Terms: conditions — COVID-19; Noncommunicable Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Comparators: Comparators without medical history of acute infection by SARS-CoV-2.
  Interventions: Other: Blood samples; Other: Six-minute walk test, Spirometry, HRCT, Heart ultrasound, Completion of questionnaires of symptoms
- Participants with NO dysfunction: Patients fully recovered by acute COVID-19 who did not present any acute organ injury during acute infection by SARS-CoV-2.
  Interventions: Other: Blood samples; Other: Six-minute walk test, Spirometry, HRCT, Heart ultrasound, Completion of questionnaires of symptoms
- Participants with Dysfunctions: Patients who presented signs of lung, heart, and kidney dysfunction during acute infection by SARS-CoV-2.
  Interventions: Other: Blood samples; Other: Six-minute walk test, Spirometry, HRCT, Heart ultrasound, Completion of questionnaires of symptoms

INTERVENTIONS:
Other: Blood samples — Blood sampling for proteomics and transcriptomics, suPAR measurement & isolation and stimulation of peripheral blood mononuclear cells, eGFR, serum creatinine, cystatin c & urea
Other: Six-minute walk test, Spirometry, HRCT, Heart ultrasound, Completion of questionnaires of symptoms — Spirometry for forced expiratory volume in the first, second, total lung capacity and diffusion capacity of carbon monoxide.

SUMMARY:
More than 660 million cases of COVID-19 have been reported worldwide, with 183 million cases in the EU alone. In several people, after recovery, the effects of the first waves of COVID-19 persisted beyond the acute phase and increased the risk of chronic multiorgan symptoms and disease. Up to 70% of people affected by COVID-19 showed reduced organ function even four months or more after COVID-19 diagnosis. Such a functional decline is associated with an increased risk of the development of non-communicable diseases (NCDs). Thus, there is an essential need for a better knowledge, tools, clinical guidelines and recommendations that it will make it possible to reduce this overrepresentation of NCDs as a consequence of the post-acute phase (PAP) of COVID-19.

The overall concept underpinning "POINT" is to i) build detailed knowledge on the link between the PAP of COVID-19 caused by previous, current, and future SARS-CoV-2 variants in vaccinated and unvaccinated people, and NCDs, ii) identify robust biomarkers and build predictive tools that help early identification and management of risk of NCDs, and iii) develop guidelines and recommendations for all parts of the healthcare value chain, allowing best prevention and care acknowledging vulnerability. The investigators will focus on the NCDs affecting pulmonary, cardiovascular and renal systems.

DETAILED DESCRIPTION:
Post-acute phase of COVID and Non-communicable diseases

Following the emergence of SARS-CoV-2, more than 660 million cases of COVID-19 have been reported worldwide, with 183 million cases in the EU alone. These numbers will continue to grow even after the disease becomes endemic. In some people, after recovery, the effects of the first waves of COVID-19 persisted beyond the acute phase and increased the risk of chronic multiorgan symptoms and disease. Up to 70% of people affected by COVID-19 showed reduced organ function even four months or more after COVID-19 diagnosis. Such a functional decline is associated with an increased risk of the development of non-communicable diseases (NCDs). This is especially true for individuals aged 65 and older as the risk of NCDs increases with age.

Diseases of the pulmonary, cardiovascular, and renal systems are the three major NCDs carrying the most significant burden for the individual as well as society. Studies have documented compromised function of these 3 organ systems in the PAP of COVID-19 in 30%-70% of patients, regardless of the severity of the acute-phase. As homeostasis of these three organs depends on interorgan communication with each other, the impact of PAP of COVID-19 on one will impact the others. The added stress of the PAP of COVID-19 increases the risk of a higher incidence and/or the risk of an accelerated progression of disease.

The prevalence and socioeconomic cost of the three NCDs is already extremely high. Without a strong focus on minimmising the increased risk of incidence and accelerated progression of the NCDs as a result of the PAP of COVID-19, up to 9 million Europeans may be affected and result in an added direct attributable cost of between 19.564 € - 31.064 € per year for each person who develop an NCD.

Beyond state of the art: pulmonary, cardiovascular and renal complications after the PAP of COVID-19

Post-acute COVID-19 and pulmonary complications - Respiratory conditions have been reported as occurring twice as often after severe COVID-19 as in the general population. In a study of 135 individuals, the incidence of impaired lung diffusing capacity (DLCO) and persistent lung damage was demonstrated in 30% of patients 12 months after acute COVID-19. In another study of 142 individuals, pulmonary abnormalities were observed by CT scans in 54% of individuals a year after acute COVID-19.

Post-acute COVID-19 and cardiovascular complications - The PAP of COVID-19 is associated with an increased risk of deep vein thrombosis up to three months after COVID-19 infection, pulmonary embolism up to six months, and a bleeding event up to two months. In a registry study of 153,760 individuals with COVID-19, the 12 month period following the acute phase was characterized by an increased risk and an excess disease burden of cardiovascular diseases, including heart failure, dysrhythmias and stroke. The risks were evident regardless of age, race, sex, and other cardiovascular risk factors. MRI revealed cardiac impairment in 78% of 100 individuals in the PAP of COVID-19.

Post-acute COVID-19 and renal complications - A study of 1733 individuals documented reduced renal function in 35% 6 months after the acute phase of COVID-19 and 13% of patients who did not have acute kidney injury (AKI) during the acute phase showed a disproportionate reduction in renal function during follow-up. A study including >89,000 individuals revealed an increased risk of adverse renal outcomes in the PAP of COVID-19.

The main unmet needs requiring action at the European level There is an urgent need to enable a better understanding of the causality between PAP of COVID-19 and the increased risk of pulmonary, cardiovascular, and renal complications and thereby an increased risk of onset of disease or aggravation of existing disease. Even though recent studies suggest such a link, there is a need for a more nuanced study of the correlation on much larger cohorts to determine the incidence and risk ratio more accurately. Furthermore, there is a need to compare the outcomes between the early, present, and potential future strains of SARS-CoV-2 variants responsible for the disease. An increased cohort size will also allow a better understanding of the impact of socioeconomic status, difference between sexes, the compounding effects of genotype, pre-existing comorbidities, and use of prescription drugs and of differences between the PAP of early strains of SARS-CoV-2 in mostly unvaccinated individuals compared with current strains in mostly vaccinated people. As this knowledge is currently incomplete, there is an immediate risk that a large part of the European population will not receive optimal and timely care.

Thus far, investigators have concluded that the functional decline of organs caused by COVID-19 cannot be explained by known risk factors. A review of the recent literature suggests that the PAP of COVID-19 is associated with immune dysregulation, elevated levels of autoantibodies, microbiota disruption and clotting and endothelial abnormalities. However, the same review also concludes that the current understanding is not sufficient to improve outcomes and calls for additional research. This underscores the involvement of unidentified molecular mechanisms responsible for the aetiology. A lack of understanding of these inhibits the development of effective biomarkers and drug candidates that allow optimal prediction of the prognosis and treatment of patients following resolution of the initial symptoms of COVID-19.

There is an urgent need for updated clinical practice guidelines and new tools to diagnose and prevent the development and aggravation of NCDs caused by the PAP of COVID-19. Currently, there are very few clinical guidelines and recommendations related to the PAP of COVID-19 and NCDs in general, and there are even fewer clinical guidelines and recommendations that focus on the effects of the PAP of COVID-19 on pulmonary, cardiovascular, and renal health. Modern clinical practice guidelines and recommendations that efficiently bridge the gap between research and current practice are invaluable for securing best quality of care, patient outcomes and cost effectiveness. Unfortunately, the development of a guideline or a recommendation does not necessarily lead to changes in clinical practice. Clinical guidelines and recommendations are not always followed, and it is estimated that approximately 30%-40% of patients receive treatment that is not based on scientific evidence and 20%-25% receive treatments that are not needed or potentially harmful.

ELIGIBILITY:
Inclusion Criteria:

Group A (comparators)

1. Adults (18 years or more) of both genders
2. Negative history of acute COVID-19

Group B (patients with ΝΟ dysfunction)

1. Adults (18 years or more) of both genders
2. History of acute COVID-19 hospitalized or non-hospitalized. All cases appearing from start of the pandemic until the last six months may apply
3. Absence of any current overt organ dysfunction
4. Absence of signs of any organ dysfunction during acute COVID-19

Group C (patients with dysfunctions)

1. Adults (18 years or more) of both genders
2. History of acute COVID-19 hospitalized or non-hospitalized. All cases appearing from start of the pandemic until the last six months may apply
3. Presence of signs of organ dysfunction of the lung, the kidneys or the heart during acute COVID-19

Exclusion Criteria:

Group A (comparators)

1. Any other co-existing disorder generating clinical symptoms
2. Failure to thrive according to the attending physicians
3. Pregnancy or lactation

Group B (patients with ΝΟ dysfunction)

1. Any other co-existing disorder generating clinical symptoms
2. Failure to thrive according to the attending physicians
3. Pregnancy or lactation

Group C (patients with dysfunctions)

1. Any other co-existing disorder generating clinical symptoms
2. Medical history of any of:

   * stage III or IV chronic obstructive pulmonary disease according to the GOLD criteria
   * pulmonary fibrosis or pulmonary hypertension
   * stage IV solid tumour malignancy under chemotherapy or radiotherapy
   * systemic sclerosis
   * congestive heart failure
   * stage II, III or IV dyspnoea according to the New York Heart Association classification before the acute COVID-19
3. Limited chance of survival for at least six months due to co-existing comorbidity(-ies) according to the judgement of the attending physicians
4. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: POINT will include patients who have participated in the studies ESCAPE, SAVE, SAVE-MORE and SAVE-LONG. For these patients blood samples and clinical data are already available (Baseline - Year 0 from ESCAPE, SAVE & SAVE-MORE and Year 1 from SAVE-LONG).
  POINT needs to enroll three groups of patients (selected by the existing biobank mentioned above, based on the inclusion and exclusion study criteria) to cover the magnitude of the spectrum of COVID-19:
  * Group A (115 Comparators): Comparators without medical history of acute infection by SARS-CoV-2.
  * Group B (115 with NO dysfunction): Patients fully recovered by acute COVID-19 who did not present any acute organ injury during acute infection by SARS-CoV-2.
  * Group C (115 with Dysfunctions): Patients who presented signs of lung, heart, and kidney dysfunction during acute infection by SARS-CoV-2.
Sampling Method: Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of any organ dysfunction during the first 48 months among patients of group C compared to group B | From enrollment to Month 48
  This is a composite endpoint which includes the development of chronic failures of at least one of lung, heart and/or kidneys

SECONDARY OUTCOMES:
The incidence of any organ dysfunction during the first 48 months among patients of group C compared to group A. | From enrollment to Month 48.
  This is a composite endpoint which includes the development of chronic failures of at least one of lung, heart and/or kidneys.
The incidence of any organ dysfunction during the first 48 months among patients of group B compared to group A. | From enrollment to Month 48.
  This is a composite endpoint which includes the development of chronic failures of at least one of lung, heart and/or kidneys.
The incidence of chronic lung failure during the first 48 months among patients of group C compared to group B. | From enrollment to Month 48.
• The incidence of chronic heart failure during the first 48 months among patients of group C compared to group B. | From enrollment to Month 48.
• The incidence of chronic renal disease during the first 48 months among patients of group C compared to group B. | From enrollment to Month 48.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Evangelos Giamarellos-Bourboulis, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (6):
- Greece (6):
  - 10th Department of Pulmonary Medicine, Sotiria Athens Hospital of Chest Diseases, Athens
  - 4th Department of Internal Medicine, ATTIKON University General Hospital, Athens
  - Obstructive Diseases Clinic, Sotiria Athens Hospital of Chest Diseases, Athens
  - Out-patient department of Infectious Diseases, Sotiria Athens Hospital of Chest Diseases, Athens
  - 1st Department of Internal Medicine, Thriasio General Hospital of Elefsina, Elefsina
  - 2nd Department of Internal Medicine, Thriasio General Hospital of Elefsina, Elefsina